CLINICAL TRIAL: NCT04176536
Title: Pharmacokinetics, Safety and Tolerability After Single Dose Administration of BI 764198 in Subjects With Moderate and Severe Renal Impairment in Comparison to Subjects With Normal Renal Function (a Mono-centric, Open-label Study With Matched-pair Design)
Brief Title: A Study in People With Normal Kidney Function and People With Reduced Kidney Function to Test How BI 764198 is Processed in the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1434-0002; 2019-003744-69 (EudraCT Number)
Record Dates: First submitted 2019-11-22; First posted 2019-11-25 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Healthy; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- All participants (Experimental)
  Interventions: Drug: BI 764198

INTERVENTIONS:
Drug: BI 764198 — Capsules

SUMMARY:
The main objective of this trial is to investigate the influence of moderate and severe renal impairment on the pharmacokinetics of a single dose of BI 764198 in comparison to a group of matched controls with normal renal function.

ELIGIBILITY:
Inclusion criteria:

* Despite of moderate and severe renal impairment (Group 1 and Group 2) male or female subjects (at least 25% of each gender) according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Estimated Glomerular filtration rate (eGFR) based on Chronic kidney disease (CKD)-EPI formula for Group 1 between 30 and 59 mL/min/1.73m², for Group 2 between 15 and 29 mL/min/1.73m² and for Group 3 ≥90 mL/min/1.73m²
* Age of 18 to 79 years (inclusive)
* Body mass index (BMI) of 18.5 to 34 kg/m^2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Male subjects, or female subjects who meet any of the following criteria from at least 30 days before the first administration of trial medication until 30 days after trial completion:

  * Use of adequate contraception, e.g. any of the following methods plus condom: implants, injectables, combined oral or vaginal contraceptives, intrauterine device
  * Sexually abstinent (defined as refraining from heterosexual intercourse during the entire period of risk)
  * A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
* Surgically sterilised (including hysterectomy)

  -- Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with levels of Follicle-stimulation hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory) Control subjects (Group 3)
* Subjects who can be matched to renal impaired subjects from Group 1 and/or Group 2 based on gender, race, age (within ±10%) and BMI (within ±10%)

Exclusion criteria:

Control subjects:

* Any finding in the medical examination (including Blood pressure (BP), Pulse rate (PR) or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Estimated Glomerular filtration rate (eGFR) calculated by Chronic kidney disease (CKD)-EPI formula < 90 mL/min/1.73m²

Subjects with moderate and severe renal impairment:

* Subject with significant diseases, in the opinion of the investigator, other than moderate or severe renal impairment. A significant disease is defined as a disease which is in the opinion of the investigator:

  * puts the subjects at risk by participating in the study
  * may influence the results of the study
  * may influence the subject's ability to participate in the study
  * is not in a stable condition Diabetic or hypertensive subjects can be entered in this trial if the disease is not significant according to those criteria.
* Moderate and severe concurrent liver function impairment (e.g. due to hepatorenal syndrome) or biliary obstruction
* Clinically relevant laboratory abnormalities (except for renal function tests or deviation of clinical laboratory values that are related to renal impairment)
* eGFR calculated by CKD-EPI formula ≥60 mL/min/1.73m² and < 30 mL/min/1.73m² for Group 1 and ≥30 mL/min/1.73m² and < 15 mL/min/1.73m² for Group 2

For all subjects:

* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 30 days of planned administration of investigational drug in the current trial, or longer if required by local regulation, or within 5 half-lives of the investigational agent taken (whichever is longer) or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 20 g per day for females and 30 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males or repeatedly greater than 470 ms in females) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

Female subjects will not be allowed to participate, if any of the following apply:

* Positive pregnancy test, pregnancy, or plans to become pregnant within 30 days after study completion
* Lactation

Male subjects will not be allowed to participate, if any of the following apply:

* Male subjects with WOCBP partner who are unwilling to use male contraception (condom or sexual abstinence) from the first administration of trial medication until 30 days after last administration of trial medication
* positive test indicating an ongoing infection with SARS-CoV-2 and clinical symptoms suggestive of the disease

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | Up to 96 hours
Cmax (maximum measured concentration of the analyte in plasma) | Up to 96 hours

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 the last quantifiable data point) | Up to 96 hours

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Kiel GmbH, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- [Derived] Schultz A, Halabi A, Seitz F, Lemmens K, Wulfrath HS, Lobmeyer MT, Retlich S, Choi W, Soleymanlou N. Phase 1 trials of BI 764198, a transient receptor potential channel 6 inhibitor, in healthy volunteers and participants with kidney impairment. Expert Opin Investig Drugs. 2025 May;34(5):415-423. doi: 10.1080/13543784.2025.2510673. Epub 2025 Jun 8. PMID 40455255
- See also: Related Info — https://www.mystudywindow.com